CLINICAL TRIAL: NCT05009667
Title: A Prospective, Multi-center Clinical Trial for Evaluating the Effectiveness and Safety of Coronary Angiography-Derived Index of Microcirculatory Resistance Measured Online by a Coronary Functional Measurement System
Brief Title: A Prospective, Multi-center Clinical Trial for Evaluating the Effectiveness and Safety of Online Coronary Angiography-Derived Index of Microcirculatory Resistance (caIMR)
Acronym: Flash III
Status: Completed | Type: Observational
Sponsor: Ge Junbo (Other)
Collaborators: RainMed Medical Group (Industry)
Responsible Party: Sponsor-Investigator, Ge Junbo, Coordinating Investigator, Fudan University
Organization: Fudan University (Other)
Other Study IDs: Flash III
Record Dates: First submitted 2021-07-23; First posted 2021-08-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Coronary Microvascular Dysfunction
Keywords: Hemodynamics; Computational fluid dynamics; Index of microcirculatory resistance; Fractional flow reserve; Angiography-derived IMR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMR first group: In this group, IMR based on pressure wire and arterial physiological detector will be measured first, and then caIMR base on angiography images and pressure sensor will be measured secondly.
  Interventions: Device: Angiography-derived Index of Microcirculatory Resistance; Device: Pressure wire-based Index of Microcirculatory Resistance
- caIMR first group: In this group, caIMR based on angiography images and pressure sensor will be measured first, and then IMR based on pressure wire and arterial physiological detector will be measured secondly.
  Interventions: Device: Angiography-derived Index of Microcirculatory Resistance; Device: Pressure wire-based Index of Microcirculatory Resistance

INTERVENTIONS:
Device: Angiography-derived Index of Microcirculatory Resistance — caIMR will be measured by pressure sensors which are produced by Suzhou Rainmed Medical Technology Co., Ltd.
  caIMR is calculated based on angiography images and Hyperemic Pa estimated from resting Pa according to prespecified equation.
Device: Pressure wire-based Index of Microcirculatory Resistance — IMR will be measured by thermodilution method with pressure wire and arterial physiological detector which are produced by St. Jude Medical.
  IMR = Pd ∙Tmn

SUMMARY:
More than 50% of patients with stable or unstable angina pectoris have no obstructive coronary arteries by angiographic visual estimation, in which coronary microvascular dysfunction (CMD) is one of the causes of myocardial ischemia and chest pain. A coronary angiography-derived index of microcirculatory resistance (caIMR) is proposed for physiological assessment of microvascular diseases in coronary circulation. The aim of the trial is to assess diagnostic performance of caIMR, using wire-derived index of microcirculatory resistance (IMR) as the reference standard.

DETAILED DESCRIPTION:
More than 50% of patients with stable or unstable angina pectoris have no obstructive coronary arteries by angiographic visual estimation, in which coronary microvascular dysfunction (CMD) is one of the causes of myocardial ischemia and chest pain. Presently, the index of microcirculatory resistance (IMR) measured by the pressure wire is recognized as standard for evaluating coronary microcirculatory function. A coronary angiography-derived index of microcirculatory resistance (caIMR) is proposed for physiological assessment of microvascular diseases in coronary circulation without pressure wire, hyperemic agents, or thermodilution method.

This study is a prospective, multi-center clinical trial. In the study, IMR (measured by pressure wire) will be used as a reference standard to evaluate the feasibility, accuracy and safety of caIMR measured by a non-invasive diagnosis system (FM21a) based on angiography images and aortic pressure wave. 116 patients eligible for inclusion criteria will be enrolled in the study. Both IMR and caIMR measurement will be performed in the same patient in a random order after angiography. The definitions of IMR and caIMR for coronary microcirculatory ischemia are IMR≥25 and caIMR≥25. The primary endpoint is the diagnostic accuracy of caIMR. The secondary endpoint is caIMR's sensitivity, specificity, positive predictive value, negative predictive value, ROC curve and AUC of caIMR diagnosis, and the diagnostic characteristics of caIMR at the vascular level.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and above, 80 years old and below, with no gender limitation;
2. Patients with stable or unstable angina or suspected myocardial ischemia;
3. Patients voluntarily participated in this clinical trial and signed an informed consent form;
4. Target coronary with <50% diameter stenosis (DS%) by visual estimation.

Exclusion Criteria:

1. Patients with suspected acute myocardial infarction;
2. Patients with old myocardial infarction;
3. Patients with primary or secondary cardiomyopathy;
4. Patients with primary or secondary heart valve disease;
5. Patients with severe cardiac insufficiency and LVEF≤35%;
6. Patients with renal insufficiency (eGFR<60ml/min (1.73m^2)) or patients undergoing dialysis;
7. Patients who are allergic to iodine contrast agents, adenosine, and ATP;
8. Patients with severe organ disease or life expectancy less than 24 months;
9. Patients who are participating in other clinical studies of investigational drugs or devices and have not reached their primary endpoint;
10. The patient who has other conditions that are not suitable for clinical trials;
11. Patients with coronary artery involved in coronary fistula and myocardial bridge;
12. The contrast media is not filled, the blood vessels are overlapped, or the target blood vessel is severely distorted, and the lesion location cannot be fully exposed, or the image quality is poor and cannot be recognized;
13. Left main coronary artery disease and right coronary artery orifice disease;
14. After angiography, the investigator believes that the patient cannot tolerate any of the detection methods between caIMR and IMR;
15. The investigator believes that the patient is not suitable for clinical trials after angiography;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable or unstable angina, or suspected myocardial ischemia.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | Through study completion, an average of 7 months.
  To compare diagnostic accuracy of caIMR for coronary microvascular dysfunction with IMR as control.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value, and negative predictive value | Through study completion, an average of 7 months.
  To compare the diagnostic performance between caIMR and IMR in the patient level, with IMR as the reference standard.
ROC curve, and AUC | Through study completion, an average of 7 months.
  Using IMR as reference standard, draw the ROC curve of caIMR. The definition of ischemia is IMR≥25.
Diagnostic performance on the vessel level | Through study completion, an average of 7 months.
  The diagnostic features of caIMR compared with IMR on the vessel level.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, PHD, Study Director — Fudan University
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Zhongnan Hospital Of Wuhan Uniersity, Wuhan, Hubei
  - Zhongshan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li J, Gong Y, Wang W, Yang Q, Liu B, Lu Y, Xu Y, Huo Y, Yi T, Liu J, Li Y, Xu S, Zhao L, Ali ZA, Huo Y. Accuracy of computational pressure-fluid dynamics applied to coronary angiography to derive fractional flow reserve: FLASH FFR. Cardiovasc Res. 2020 Jun 1;116(7):1349-1356. doi: 10.1093/cvr/cvz289. PMID 31693092
- [Background] Fearon WF, Balsam LB, Farouque HM, Caffarelli AD, Robbins RC, Fitzgerald PJ, Yock PG, Yeung AC. Novel index for invasively assessing the coronary microcirculation. Circulation. 2003 Jul 1;107(25):3129-32. doi: 10.1161/01.CIR.0000080700.98607.D1. Epub 2003 Jun 23. PMID 12821539
- [Background] Ford TJ, Berry C. How to Diagnose and Manage Angina Without Obstructive Coronary Artery Disease: Lessons from the British Heart Foundation CorMicA Trial. Interv Cardiol. 2019 May 21;14(2):76-82. doi: 10.15420/icr.2019.04.R1. eCollection 2019 May. PMID 31178933
- [Background] Kunadian V, Chieffo A, Camici PG, Berry C, Escaned J, Maas AHEM, Prescott E, Karam N, Appelman Y, Fraccaro C, Louise Buchanan G, Manzo-Silberman S, Al-Lamee R, Regar E, Lansky A, Abbott JD, Badimon L, Duncker DJ, Mehran R, Capodanno D, Baumbach A. An EAPCI Expert Consensus Document on Ischaemia with Non-Obstructive Coronary Arteries in Collaboration with European Society of Cardiology Working Group on Coronary Pathophysiology & Microcirculation Endorsed by Coronary Vasomotor Disorders International Study Group. Eur Heart J. 2020 Oct 1;41(37):3504-3520. doi: 10.1093/eurheartj/ehaa503. PMID 32626906
- [Background] Fearon WF, Farouque HM, Balsam LB, Caffarelli AD, Cooke DT, Robbins RC, Fitzgerald PJ, Yeung AC, Yock PG. Comparison of coronary thermodilution and Doppler velocity for assessing coronary flow reserve. Circulation. 2003 Nov 4;108(18):2198-200. doi: 10.1161/01.CIR.0000099521.31396.9D. Epub 2003 Oct 20. PMID 14568891
- [Background] Ai H, Feng Y, Gong Y, Zheng B, Jin Q, Zhang HP, Sun F, Li J, Chen Y, Huo Y, Huo Y. Coronary Angiography-Derived Index of Microvascular Resistance. Front Physiol. 2020 Dec 16;11:605356. doi: 10.3389/fphys.2020.605356. eCollection 2020. PMID 33391020
- [Background] Aarnoudse W, Fearon WF, Manoharan G, Geven M, van de Vosse F, Rutten M, De Bruyne B, Pijls NH. Epicardial stenosis severity does not affect minimal microcirculatory resistance. Circulation. 2004 Oct 12;110(15):2137-42. doi: 10.1161/01.CIR.0000143893.18451.0E. Epub 2004 Oct 4. PMID 15466646
- [Background] Kobayashi Y, Lee JM, Fearon WF, Lee JH, Nishi T, Choi DH, Zimmermann FM, Jung JH, Lee HJ, Doh JH, Nam CW, Shin ES, Koo BK. Three-Vessel Assessment of Coronary Microvascular Dysfunction in Patients With Clinical Suspicion of Ischemia: Prospective Observational Study With the Index of Microcirculatory Resistance. Circ Cardiovasc Interv. 2017 Nov;10(11):e005445. doi: 10.1161/CIRCINTERVENTIONS.117.005445. PMID 29146670
- [Background] Yoon MH, Tahk SJ, Yang HM, Woo SI, Lim HS, Kang SJ, Choi BJ, Choi SY, Hwang GS, Shin JH. Comparison of accuracy in the prediction of left ventricular wall motion changes between invasively assessed microvascular integrity indexes and fluorine-18 fluorodeoxyglucose positron emission tomography in patients with ST-elevation myocardial infarction. Am J Cardiol. 2008 Jul 15;102(2):129-34. doi: 10.1016/j.amjcard.2008.03.024. Epub 2008 May 29. PMID 18602508
- [Background] Williams RP, de Waard GA, De Silva K, Lumley M, Asrress K, Arri S, Ellis H, Mir A, Clapp B, Chiribiri A, Plein S, Teunissen PF, Hollander MR, Marber M, Redwood S, van Royen N, Perera D. Doppler Versus Thermodilution-Derived Coronary Microvascular Resistance to Predict Coronary Microvascular Dysfunction in Patients With Acute Myocardial Infarction or Stable Angina Pectoris. Am J Cardiol. 2018 Jan 1;121(1):1-8. doi: 10.1016/j.amjcard.2017.09.012. Epub 2017 Oct 10. PMID 29132649
- [Background] De Maria GL, Alkhalil M, Wolfrum M, Fahrni G, Borlotti A, Gaughran L, Dawkins S, Langrish JP, Lucking AJ, Choudhury RP, Porto I, Crea F, Dall'Armellina E, Channon KM, Kharbanda RK, Banning AP. Index of Microcirculatory Resistance as a Tool to Characterize Microvascular Obstruction and to Predict Infarct Size Regression in Patients With STEMI Undergoing Primary PCI. JACC Cardiovasc Imaging. 2019 May;12(5):837-848. doi: 10.1016/j.jcmg.2018.02.018. Epub 2018 Apr 18. PMID 29680355
- [Derived] Huang D, Gong Y, Fan Y, Zheng B, Lu Z, Li J, Huo Y, Escaned J, Huo Y, Ge J. Coronary angiography-derived index for assessing microcirculatory resistance in patients with non-obstructed vessels: The FLASH IMR study. Am Heart J. 2023 Sep;263:56-63. doi: 10.1016/j.ahj.2023.03.016. Epub 2023 Apr 12. PMID 37054908